CLINICAL TRIAL: NCT01883661
Title: Role of Autologous Bone Marrow Derived Mono Nuclear Stem Cell (MNCs) In Patient With Multiple Sclerosis .It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of BMMNC in Multiple Sclerosis (MS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Sub Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BM/2013/MS/01
Record Dates: First submitted 2013-06-12; First posted 2013-06-21 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Sclerosis
Keywords: stem cell; Multiple Sclerosis; BMMNC
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMMNC (Other): Administration of of Bone Marrow derived Mono Nuclear Stem Cell (MNCs)
  Interventions: Biological: BMMNC

INTERVENTIONS:
Biological: BMMNC — Bone Marrow derived Mono Nuclear Stem Cell (MNCs) by intravenously route total 3 doses in one month period .

SUMMARY:
The aim of this study is to prove the BMMNC Therapy in Multiple sclerosis, and to control symptoms and help to maintain a normal quality of life of suffering patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is considered to be an autoimmune disease that is caused by the immune system attacking the central nervous system (CNS) leading to myelin loss and axonal damage, resulting in long-term disability. The pathophysiology of MS is complex with involvement of genetic and environmental factors that define the susceptibility to generate the autoimmune attack. MS is caused by damage to the myelin sheath, the protective covering that surrounds nerve cells. When this nerve covering is damaged, nerve signals slow down or stop.The nerve damage is caused by inflammation. Inflammation occurs when the body's own immune cells attack the nervous system. Currently, treatment of MS relays mainly on immunosuppression combined with monoclonal antibodies and steroid therapies.The most advanced application for MSCs in the neurological clinical arena is in multiple sclerosis.This clinical study time period is for 1 year. This study is carried out to see the role of BMMNC cell Therapy in Multiple sclerosis, and to control symptoms and help to maintain a normal quality of life of suffering patients.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Diagnosis of MS, Aged 18 - 65 years. Duration of disease: >5 years Signed, written informed consent Willing and able to comply with study visits according to protocol for the full study period

Exclusion Criteria:

* Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to interpret the results
* Patient with any active or chronic infection
* No life-threatening organ dysfunction.
* Pregnancy or risk of pregnancy.
* Patients who are seropositive for HIV1, HIV2, Hepatitis B Surface Antigen, and Hepatitis C
* Patients unable to give written informed consent in accordance with research ethics board guidelines
* Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
* Treatment with interferon-beta or glatiramer acetate within the 30 days prior to randomization
* Treatment with corticosteroids within the 30 days prior to randomization
* Current treatment with an investigational therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
analysis of patients symptoms | baseline and 6 months
  Improvement in patients symptoms

SECONDARY OUTCOMES:
changes in Expanded Kurtzke Disability Status Score scale | baseline and 6 months
  The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis.the evaluation will be done after 6 month
changes in clinical variables | baseline and 6 months
Quality Of life questionnaire | baseline and 6 months
changes in MRI scan report | baseline and 6 months
changes in cerebrospinal fluid tests | baseline and 6 months
Changes in analysis of visual evoked potential test | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India